CLINICAL TRIAL: NCT05258708
Title: Predictive Value of Reactogenicity for Anti-SARS-CoV-2 Antibody Response in mRNA-1273 Recipients: a Multicenter Prospective Cohort Study
Brief Title: COVID-19 Vaccine Reactogenicity and Immunogenicity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Catholic Kwandong University (Other); Ajou University School of Medicine (Other); Hallym University Kangnam Sacred Heart Hospital (Other); Korea University Anam Hospital (Other); Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Joon Young Song, MD, PhD, Korea University Guro Hospital
Other Study IDs: 2021GR0274
Record Dates: First submitted 2022-02-25; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Vaccine Immune Response; Vaccine Adverse Reaction
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Biological: mRNA-1273 COVID-19 vaccine — two doses of mRNA-1273 vaccine at 28-day intervals

SUMMARY:
Analysis of antibody kinetics after vaccination with mRNA-1273 and factors influencing the vaccine immunogenicity

DETAILED DESCRIPTION:
We conducted a prospective study on healthy young adults who were to receive two doses of mRNA-1273 vaccine at 28-day intervals. After each dose, adverse events were prospectively evaluated, and blood samples were collected. The correlation between humoral immune response and reactogenicity after vaccination was determined. In addition, long-term anti-SARS-CoV-2 antibody kinetics will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* who were willing to receive the mRNA-1273 vaccine

Exclusion Criteria:

* previously diagnosed with laboratory-confirmed COVID-19
* history of autoimmune disease
* immunocompromised, pregnant, or breastfeeding

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adults between the ages of 19 and 55 years who were willing to receive the mRNA-1273 vaccine were enrolled in the study and provided written informed consent
Sampling Method: Probability Sample
Enrollment: 179 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
The correlation between humoral immune response and reactogenicity after vaccination | The correlation between reactogenicity after dose 1 and immunogenicity at T1 (28 days after dose 1 prior to the 2nd dose) and T2 (28 days after dose 2); the correlation between reactogenicity after vaccine dose 2 and immunogenicity at T2
  The correlation between humoral immune response and reactogenicity after vaccination

SECONDARY OUTCOMES:
anti-SARS-CoV-2 antibody | before vaccination (T0), 28 days after the first dose prior to the second dose (T1), and 28 days after the second dose (T2)
  SARS-CoV-2 immunoglobulin G (IgG) assay (Abbott Laboratories, Chicago, IL, USA)
neutralizing antibody titer | before vaccination (T0), 28 days after the first dose prior to the second dose (T1), and 28 days after the second dose (T2)
  plaque reduction neutralization test was performed using wild-type SARS-CoV-2 virus (BetaCoV/Korea/KCDC03/2020)
reactogenicity after vaccination | Seven days after each dose of vaccine
  record the occurrence, severity, and duration of solicited AEs using a standardized electronic questionnaire
Long-term persistence of anti-SARS-CoV-2 antibody and neutralizing antibody titer | At 3 months and 6 months after dose 1
  SARS-CoV-2 immunoglobulin G (IgG) assay (Abbott Laboratories, Chicago, IL, USA); plaque reduction neutralization test was performed using wild-type SARS-CoV-2 virus (BetaCoV/Korea/KCDC03/2020)

CONTACTS AND LOCATIONS:
Overall Officials: Joon Young Song, Principal Investigator — Korea University Guro Hospital
Locations (5):
- South Korea (5):
  - Catholic Kwandong University, Incheon
  - Kangnam Sacred Heart Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, International St. Mary's Hospital, Gangnam Sacred Heart Hospital, Ajou University School of Medicine, Korea University Anam Hospital, Seoul
  - Ajou University School of Medicine Hallym University, Suwon

IPD SHARING:
Plan to Share IPD: Undecided
We will make a decision after discussion with the staff of other hospitals. We will share data on adverse events and immunogenicity.